CLINICAL TRIAL: NCT05964244
Title: Evaluate the Impact of Noninvasive (NIV) With Expiratory Washout on Respiratory Rate of Patients With Acute Hypercapnic Respiratory Failure. A Prospective, Randomized Cross Over Pilot Investigation.
Brief Title: Impact of Noninvasive With Expiratory Washout on Respiratory Rate of Patients With Acute Hypercapnic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FisherPaykel
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Crossover study where each participant receives NIV on the Vela investigational mask and the Nivairo standard mask for one hour each in random order.
Who Masked: Outcomes Assessor
Masking Description: NIV masks can not be masked during the treatments. Only the analysis will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Noninvasive ventilation (CPAP or bilevel) with the Vela investigational mask for 1 hour (Experimental): Pressure settings for noninvasive ventilation to be set as required to provide optimal respiratory support for each patient. Not to be changed during the 2 hours of the study.
  Interventions: Device: Vela Investigational Mask
- Noninvasive ventilation (CPAP or bilevel) with the standard mask (Nivairo) for 1 hour (Active Comparator): Pressure settings for noninvasive ventilation to be set as required to provide optimal respiratory support for each patient. Not to be changed during the 2 hours of the study.
  Interventions: Device: Nivairo Standard Mask

INTERVENTIONS:
Device: Vela Investigational Mask — Wear mask to enable the delivery of noninvasive ventilation (CPAP or bilevel) therapy.
  Arms: Noninvasive ventilation (CPAP or bilevel) with the Vela investigational mask for 1 hour
Device: Nivairo Standard Mask — Wear mask to enable the delivery of noninvasive ventilation (CPAP or bilevel) therapy.
  Arms: Noninvasive ventilation (CPAP or bilevel) with the standard mask (Nivairo) for 1 hour

SUMMARY:
This study will determine if NIV using the Vela investigational mask with expiratory washout of the upper airway more effectively reduces respiratory rate in acute patients with hypercapnic respiratory failure. Patients admitted to hospital with acute respiratory failure (ARF) will be assessed for hypercapnic ARF by normal hospital protocols. Patients requiring noninvasive ventilation (NIV) will be set up on NIV as prescribed per standard of care. Enrollment onto the investigation will occur after the patient has been allowed to stabilize on NIV . Patients that meet the inclusion/exclusion criteria will be approached for consent. Investigation participants will receive two masks in random order;

1. NIV for one hour with the investigational mask (Vela)
2. NIV for one hour with the standard mask (Nivairo).

Participants will have their physiological respiratory parameters recorded.

DETAILED DESCRIPTION:
This is a simple study. Patients who are already on noninvasive ventilation (NIV) for acute respiratory failure will be approached for the study within the first 24 hours on NIV therapy.

The study will be conducted as described above. After the study patients will be able to choose which mask they continue their NIV on. They will continue NIV as part of their normal hospital care.

ELIGIBILITY:
Inclusion Criteria:

* Have type II acute respiratory failure (ARF) and have been prescribed NIV
* Arterial blood gas (ABG) Partial pressure of arterial carbon dioxide greater or equal to 6.0 kilopascals (45 millimeters of mercury)
* Arterial blood gas acidity greater or equal to 7.35 prior to bilevel commencement
* On NIV for 24 hours or less
* Negative Covid-19 test
* Are 18 years or older

Exclusion Criteria:

* Contraindicated for NIV
* On NIV in Emergency Department/ ward for more than 24 hours, within the last 48 hours
* NIV is likely to fail and/or intubation be required, at the doctor's discretion
* CPAP or bilevel pressure of 25 centimeters of water or more is required
* Unable to tolerate NIV for the duration of the investigation
* Do not fit the investigational mask or the standard mask
* Pregnancy (tested under standard care)
* Agitated
* Unable to understand the consent process

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in respiratory rate | 1 hour
  The change in patient's respiratory rate over the 1 hour of the study arm

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.